CLINICAL TRIAL: NCT04428268
Title: Phase II, Randomized, Double-blind, Controlled Clinical Trial Evaluating the Efficacy and Safety of Chloroquine + Low Dose Losartan Compared to Chloroquine Monotherapy in Subjects With SARS-CoV-2 Pneumonia
Brief Title: Chloroquine + Losartan Compared to Chloroquine Alone for the Treatment of COVID-19 Pneumonia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: evidence showed chloroquine is not effective against COVID-19
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. Adrian Camacho-Ortiz, Head of the Infectious Disease Department, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IF20-00003
Record Dates: First submitted 2020-04-26; First posted 2020-06-11 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; SARS-CoV-2 pneumonia; Chloroquine phosphate; Losartan
MeSH Terms: conditions — COVID-19 | interventions — chloroquine diphosphate; Losartan

STUDY DESIGN:
Intervention Model Description: double blind randomized clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: investigator will not be aware of the treatments or outcomes until the end of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chloroquine (Active Comparator): Patients will receive chloroquine phosphate 450 mg every 12 hours orally
  Interventions: Drug: Chloroquine Phosphate Tablets
- Chloroquine plus losartan (Experimental): Patients will receive Chloroquine phosphate 450mg orally every 12hrs plus Losartan 25mg orally every 12hrs
  Interventions: Drug: Chloroquine Phosphate Tablets

INTERVENTIONS:
Drug: Chloroquine Phosphate Tablets — Orally administered
  Other Names: Losartan tablets

SUMMARY:
Study design Phase 2, double blinded, single-center, 1:1 randomized clinical trial of Chloroquine vs Chloroquine/losartan for the treatment of SARS-CoV-2 pneumonia in non-critically ill subjects

DETAILED DESCRIPTION:
Study design Phase 2, blinded, single-center, 1: 1 randomized clinical trial for the treatment of SARS-CoV-2 pneumonia in non-critically ill subjects. Two of the co-investigators and the data analyst will remain blind to group allocation until after statistical analysis.

The groups will consist of subjects receiving in one arm PO Chloroquine 450mg every 12 hours and in the other arm, in addition to chloroquine, PO Losartan 25mg every 24 hours. Study drugs will be administered for a total of 10 days enterally.

Baseline demographics and clinical characteristics will be registered and periodically during the study.

nasopharyngeal swabs will be taken every 48hrs during hospitalization to determine the presences and viral load of SARS-CoV-2, and daily EKG for QT interval monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥18 years.
2. Oral tolerance or access for enteral administration of medication.
3. PCR or IgM for SARS-CoV-2 positive.
4. Negative pregnancy test in case of a woman of reproductive age.
5. Signature of a document proving informed consent.
6. Hospital admission for SARS-CoV-2 pneumonia.

Exclusion Criteria:

1. New alteration of the state of alert that does not revert after interventions 60 minutes after hospital admission.
2. Mean Arterial Pressure (MAP) ≤ 65mmHg despite initial resuscitation on arrival at the centre.
3. History of allergy to chloroquine, hydroxychloroquine, piperaquine or primaquine.
4. Known patient with hearing loss.
5. Received chloroquine or hydroxychloroquine in the last 3 months.
6. Patients with cirrhosis or elevation of aspartate transaminase (AST) or alanine transaminase (ALT) greater than three times the upper normal limit.
7. Patients with calculated glomerular filtration rate by Modification of Diet in Renal Disease study equation (MDRD) < 30ml/min 1.73 m2.
8. Patients known to be deficient in 6-phosphate dehydrogenase
9. Patients known to have retinopathy or macular disease.
10. History of acute myocardial infarction in the last 6 months, unstable angina, ventricular tachycardia, ventricular fibrillation or class III-IV heart failure according to New York Heart Association.
11. Electrocardiogram QTc interval ≥ 480 ms.
12. Patients with hypomagnesemia or uncorrected hypokalemia.
13. Patients with a history of psychiatric illness.
14. Patients who are pregnant or nursing.
15. Patients taking quinolones, dextropropoxyphene, amiodarone, flecainide, cisapride, domperidone, atazanavir or lopinavir.
16. Patients with acute pancreatitis.
17. Patients who the investigators deem unsuitable for participation in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Overall mortality | 28 days
  Determine all-cause mortality up to 28 days after randomization of Chloroquine Phosphate Compared to Chloroquine Phosphate plus Losartan in Non-Critically Ill Patients with SARS-CoV-2 Pneumonia.

SECONDARY OUTCOMES:
Clinical outcome assessment | 28 days
  Compare the clinical outcome of Chloroquine Phosphate treatment vs Chloroquine Phosphate plus Losartan in the follow-up visit at the end of treatment. Acording to NIH and FDA definitions
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 28 days
  Assess the adverse events associated to chloroquine and chloroquine plus losartan at 28 days
Time to negative SARS-CoV-2 test | 28 days
  Time to negative Polymerase chain reaction (PCR) test from baseline: testing every 48hrs until a negative result

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Camacho Ortiz, MD, Principal Investigator — Hospital Universitario "Dr. Jose Eleuterio Gonzalez", UANL
Locations (1):
- Hospital Universitario José E. Gonzalez, Monterrey, Nuevo León, Mexico